CLINICAL TRIAL: NCT06505954
Title: PREVALENCE OF LOWER URINARY TRACT SYMPTOMS AND CONTRIBUTING FACTORS AMONG MEDICAL STUDENTS
Brief Title: LOWER URINARY TRACT SYMPTOMS
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Muharrem Baturu, Assistant Proffesor, University of Gaziantep
Other Study IDs: GAUN-Urology-Baturu-002
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Medical students; Prevalence
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Participant who has lower urinary tract symptoms
  Interventions: Other: Survey study
- 2: Participant who doesn't have lower urinary tract symptoms

INTERVENTIONS:
Other: Survey study — Survey study among medical students about lower urinary tract symptoms
  Groups: 1

SUMMARY:
Lower urinary tract symptoms (LUTS) are observed in individuals with pathologies affecting the lower urinary system, such as detrusor overactivity, sphincter weakness, or sensory bladder disorder. LUTS can be categorized into storage, voiding, and post-micturition symptoms. Storage problems include increased frequency of urination, nocturia, urinary urgency, and incontinence. Voiding symptoms include decreased urine flow rate, hesitancy, and terminal dribbling, while post-micturition symptoms include post-micturition dribble and a sensation of incomplete bladder emptying. The prevalence of LUTS increases with age and is influenced by factors such as metabolic syndrome, gender, caffeine consumption habits, chronic psychological stress, bladder dysfunction, smoking, alcohol use, and constipation.

This study aims to investigate the prevalence of LUTS and contributing factors among medical students, a young population undergoing a stressful educational process.

A 43-question survey was prepared for all medical students from years 1 to 6. The survey included the Constipation Scoring System (CSS) to evaluate constipation, the Generalized Anxiety Disorder-7 (GAD-7) score to assess anxiety levels, and the Core Lower Urinary Tract Symptom Score (CLSS) to query LUTS. The survey also collected data on participants' dietary habits, smoking, alcohol and caffeine consumption, living conditions, age, gender, body mass index (BMI), and educational level. The study was approved by the local ethics committee of Gaziantep University (approval number 2024/234).

ELIGIBILITY:
Inclusion Criteria:

-All medical students from committee 1 to 6.

Exclusion Criteria:

* Participants who filled out the survey questions incompletely or incorrectly
* Participants who had additional diseases
* Participants who used medication for psychiatric or cardiac reasons
* Participants who had undergone surgery that could affect bladder function

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical students who have lower urinary tract symptoms are goal populations.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of lower urinary tract symptoms | Last six months

SECONDARY OUTCOMES:
Contributing factors | Last six months
  data on participants' dietary habits, smoking, alcohol and caffeine consumption, living conditions, age, gender, body mass index (BMI), and educational level,anxiety level and constipation degree will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Muharrem Baturu, Study Chair — Gaziantep University Faculty of Medicine, Department of Urology
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided